CLINICAL TRIAL: NCT00187629
Title: Phosphate Intake's Effect on the Skeletal System Calcitropic Hormones and FGF23 - Pilot Study
Brief Title: Phosphate Intake's Effect on the Skeletal System - Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: H40550-24730
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2013-10

CONDITIONS: Healthy; Kidney Failure, Chronic
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Phosphorus, Dietary

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): dietary phosphorus
  Interventions: Behavioral: dietary phosphorus
- 2 (Active Comparator): other
  Interventions: Behavioral: dietary phosphorus

INTERVENTIONS:
Behavioral: dietary phosphorus — varying amts dietary phosphorus

SUMMARY:
The purpose of this study is to determine the effects of different amounts of phosphorus in the diet on hormones that control phosphorus and bone health both in men who are healthy and in ones who have moderate kidney disease.

DETAILED DESCRIPTION:
Chronic kidney disease affects 11% of the US population; over half of those affected have skeletal manifestations of their renal disease. Renal osteodystrophy is a complex disease, in which multiple mineral systems and related hormones play a role, including phosphate homeostasis. Phosphate regulation primarily depends on renal handling of phosphate, which is partly controlled by parathyroid hormone and vitamin D. However, other mediators in this system clearly exist. Recently, evidence has been accruing that one such factor may be FGF23, a protein produced by osteogenic cells. States of excess FGF23 are associated with marked phosphate wasting, hypophosphatemia, osteomalacia, and inappropriately low calcitriol. FGF23 levels are measurable in healthy humans and markedly elevated in patients who require hemodialysis, although its physiologic role in either state is unknown. Some retrospective evidence suggests that FGF23 is affected by phosphate intake. We are performing a pilot study to gather preliminary data describing the response of FGF23 to changes in dietary phosphorus intake in healthy men and in men with moderate renal insufficiency. The specific aims of this pilot study are: 1) To examine the physiologic effects of alterations in dietary phosphorus on FGF23 in healthy subjects; 2) To examine the physiologic response of FGF23 to dietary phosphorus alterations in patients with moderate renal failure; 3) To assess whether serum levels of 1,25-dihydroxyvitamin D vary inversely with those of FGF23 when dietary phosphate is changed; 4) To determine the temporal pattern of calcitropic hormones and FGF23 in response to dietary phosphate changes; and 5) To determine the variability of the changes in serum FG 23 in response to dietary phosphate manipulations. The proposed research plan is a dietary intervention trial in which we will study the response of serum FGF23 levels to diets with varying phosphorus contents in healthy adults and adults with moderate renal insufficiency.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Men 21-65 years old with Creatinine clearance > 70 ml/min/1.73 m2 as calculated using the equation derived from the Modification of Diet in Renal Disease (MDRD) study
* Men 21-65 years old with Creatinine clearance between 30 and 59 ml/min/1.73 m2 as calculated using the equation derived from the MDRD study31

Exclusion Criteria:

* Medications affecting bone metabolism
* Abnormal liver or GI function
* Extreme electrolyte abnormalities
* BMI >30 kg/m2

Ages: 21 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2004-03; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
urine phosphorus | Daily

CONTACTS AND LOCATIONS:
Overall Officials: Diana M Antoniucci, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, California, United States